CLINICAL TRIAL: NCT04964128
Title: Evaluation of Meal Gesture Dosing in Adults With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP339
Record Dates: First submitted 2021-07-06; First posted 2021-07-15 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Type 1 Diabetes
Keywords: Advanced Hybrid Closed Loop; Meal Gesture Dosing; Klue™ Health App
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- meal gesture dosing for unannounced meals within the AHCL System (Experimental)
  Interventions: Device: MiniMed™ 780G insulin pump with Klue Health app utilizing meal gesture micro insulin dosing (meal gesture dosing)

INTERVENTIONS:
Device: MiniMed™ 780G insulin pump with Klue Health app utilizing meal gesture micro insulin dosing (meal gesture dosing) — The AHCL system with Meal Gesture Dosing evaluated in this study includes a commercial/CE-Marked insulin pump with investigational software, and the Klue Health mobile app with investigational software (installed on Apple Watch) for meal gesture detection and micro dosing.

SUMMARY:
The purpose of this feasibility study is to evaluate subject safety of using the Klue Health app utilizing meal gesture micro insulin dosing (meal gesture dosing) within the AHCL system in adult subjects with type 1 diabetes in a clinic setting.

DETAILED DESCRIPTION:
This study is a single-center, single arm study in adult subjects with type 1 diabetes utilizing AHCL System with meal gesture detection and micro dosing (meal gesture dosing). Meal gesture dosing is a mode whereby meal announcements are not entered manually by the user. Instead, when meal gesture dosing is active, meal announcements are generated automatically by the system based on the detection of eating gestures and micro doses of insulin are given.

Overall subject participation will be approximately 3 weeks to 6 months.

A total of up to 40 subjects (aged 18-75) may be enrolled at one investigational center in Israel to have at least 16 subjects complete the study.

The study consists of a run-in period and a study period. The run-in period is intended to allow subjects to become familiar with using the study pump system with the SmartGuard feature active and wearing the watch. Subjects should use the same insulin they will be using during the study period.

During the first week of the study period, subjects will undergo a 5-day at-home baseline meal challenge at specific meals on each day. The Klue app will be set to monitoring-mode. After run-in period and completion of the 5-day at-home study period with baseline meal challenges, study subjects will check into the clinic for a 5-day (4 nights) intervention. Study subjects will wear the system with Klue meal gesture dosing activated for the entire duration of the 5-day intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Is age 18-75 years at time of screening
2. Has a clinical diagnosis of type 1 diabetes for 2 years or more as determined via source documentation
3. Pump therapy for greater than 6 months prior to screening
4. Real-time continuous glucose monitoring (RT-CGM) experience greater than 3 months prior to screening
5. Must have a minimum daily insulin requirement (Total Daily Dose) of greater than or equal to 8 units
6. Is willing to perform ≥2 fingerstick blood glucose measurements daily
7. Is willing to perform required sensor calibrations
8. Is willing to wear the system continuously throughout the study
9. If subject has celiac disease, it has been adequately treated as determined by the investigator
10. If the subject has had any of the following cardiovascular events more than 1 year prior to of screening: myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, or ventricular rhythm disturbances they should be cleared by a cardiologist prior to participation, if deemed necessary by the investigator.
11. If the subject has had any of the following cardiovascular events within 1 year of screening: myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, or ventricular rhythm disturbances, they should be cleared by a cardiologist prior to participation.
12. Is of legal age and capable of providing consent
13. Is fluent in speaking, reading and understanding English

Exclusion Criteria:

1. Has a history of 1 or more episodes of severe hypoglycemia, which resulted in any the following during the 6 months prior to Screening:

   1. Medical assistance (i.e. Paramedics, Emergency Room (ER) or Hospitalization)
   2. Coma
   3. Seizures
2. Has been hospitalized or has visited the ER in the 6 months prior to Screening resulting in a primary diagnosis of uncontrolled diabetes
3. Has had Diabetic Ketoacidosis (DKA) in the 6 months prior to Screening.
4. Is unable to tolerate tape adhesive in the area of sensor placement
5. Has any unresolved adverse skin condition in the area of sensor placement (e.g., psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection)
6. Women of child-bearing potential who have a positive pregnancy test at Screening or plan to become pregnant during the course of the study
7. Women who are breastfeeding
8. Females who are sexually active and able to conceive will be excluded if they are not using an effective method of contraception and do not agree to continue using an effective method of contraception for the duration of the study as determined by investigator.
9. Is being treated for hyperthyroidism at time of Screening
10. Has a diagnosis of adrenal insufficiency
11. Is using hydroxyurea at time of screening or plans to use it during the study
12. Is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks
13. Is currently abusing illicit drugs, marijuana, alcohol or prescription drugs (other than nicotine), per investigator judgement
14. Is using pramlintide (Symlin), DPP-4 inhibitor, GLP-1 agonists (as liraglutide (Victoza or other), metformin, SGLT2 inhibitors (as canagliflozin (Invokana)) at time of screening
15. Has a history of visual impairment which would not allow subject to participate in the study and perform all study procedures safely, as determined by the investigator
16. Is diagnosed with current eating disorder such as anorexia or bulimia
17. Has been diagnosed with chronic kidney disease that results in chronic anemia
18. Is on dialysis
19. Is a member of the research staff involved with executing the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-07-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roy A, Grosman B, Benedetti A, Engheta B, Miller D, Laron-Hirsh M, Cohen Y, Re R, Edd SN, Vigersky R, Cohen O, Tirosh A. An Automated Insulin Delivery System with Automatic Meal Bolus Based on a Hand-Gesturing Algorithm. Diabetes Technol Ther. 2024 Sep;26(9):633-643. doi: 10.1089/dia.2023.0529. Epub 2024 Mar 12. PMID 38417017

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 1 studied the Klue Health app with investigational software release tag 1.0, and Phase 2 studied the Klue Health App with investigational software release tag 2.0. Both phases included Run-In and Study Periods. The participant flow numbers for each phase reflect the participation through both the run-in and study periods within the phase.
  Both phases had 18 total participants starting the phase, with 8 subjects being unique to each phase. 10 subjects participated in both Phases 1 and 2.
Groups:
- AHCL System With Meal Gesture Detection and Micro Dosing (Meal Gesture Dosing): 18-75 year old subjects with type 1 diabetes utilizing AHCL System with meal gesture detection and micro dosing (meal gesture dosing)
Period: Phase 1 (Software Release Tag 1.0)
Arm/Group | AHCL System With Meal Gesture Detection and Micro Dosing (Meal Gesture Dosing)
Started | 18 (8 subjects participated in both phases 1 and 2, and there were 10 subjects who participated in only Phase 1)
Completed | 17
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Phase 2 (Software Release Tag 2.0)
Arm/Group | AHCL System With Meal Gesture Detection and Micro Dosing (Meal Gesture Dosing)
Started | 18 (8 subjects participated in both phases 1 and 2, and there were 10 subjects who participated in only Phase 2)
Completed | 17
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Overall number of baseline participants reflects all unique subjects participating in phases 1 and 2. There were 8 subjects participating in both phases, so although there were 18 subjects in each phase, there were only 28 unique subjects in the entire study.
Arm/Group | AHCL System With Meal Gesture Detection and Micro Dosing (Meal Gesture Dosing)
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Israel | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time in Range (Phase 1, Software Release Tag 1.0)
Description: Overall mean percentage of Post-prandial Time in range (% of SG within 70-180 mg/dL) at home and In-Clinic Period during Phase 1
Time Frame: Overall subject participation lasted approximately 3 weeks to 6 months, which included a run-in period and a study period (5 days at-home and 5 days in-clinic). The time in range metrics are considered in a 4 hours window after each of the test meals.
Population: Number of participants only includes those that had data available
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- At-Home: Phase 1 studied the Klue Health app with investigational software release tag 1.0.
  This portion refers to the baseline 5-day meal challenges done at home.
- In-Clinic: Phase 1 studied the Klue Health app with investigational software release tag 1.0.
  This portion refers to the 5-day intervention done in clinic.
Arm/Group | At-Home | In-Clinic
Number analyzed (Participants) | 17 | 17
percentage of time
  Meal 1 (Large Meal with Low Carbohydrate Count): number analyzed (Participants) | 17 | 16
  Meal 1 (Large Meal with Low Carbohydrate Count) | 76.1 (28.7) | 84.3 (14.9)
  Meal 2 (Small Meal with High Carbohydrate Count) | 65.5 (35.7) | 48 (28.1)
  Meal 3 (Typical Meal Size with Medium Carbohydrate Count): number analyzed (Participants) | 17 | 16
  Meal 3 (Typical Meal Size with Medium Carbohydrate Count) | 70 (33.5) | 70.9 (27.4)
  Meal 4 (Typical Meal Size with High Carbohydrate Count): number analyzed (Participants) | 17 | 16
  Meal 4 (Typical Meal Size with High Carbohydrate Count) | 63.9 (28.8) | 27.3 (12.2)
  Meal 5 (Typical Meal Size with Low Carbohydrate Count): number analyzed (Participants) | 16 | 16
  Meal 5 (Typical Meal Size with Low Carbohydrate Count) | 82.7 (25) | 73.5 (30.5)

2. Primary Outcome: Percentage of Time in Range (Phase 2, Software Release Tag 2.0)
Description: Overall mean percentage of Post-prandial Time in range (% of SG within 70-180 mg/dL) at home and In-Clinic Period during Phase 2
Time Frame: Overall subject participation lasted approximately 3 weeks to 6 months, which included a 5 day at-home and a 5-day in-clinic period. The time in range metrics are considered in a 4 hours window after each of the test meals.
Population: Number of participants only includes those that had data available
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- At-Home: Phase 2 studied the Klue Health app with investigational software release tag 2.0.
  This portion refers to the baseline 5-day meal challenges done at home.
- In-Clinic: Phase 2 studied the Klue Health app with investigational software release tag 2.0.
  This portion refers to the 5-day intervention done in clinic.
Arm/Group | At-Home | In-Clinic
Number analyzed (Participants) | 17 | 17
percentage of time
  Meal 1 (Long Meal with Low Carbohydrate Count): number analyzed (Participants) | 16 | 16
  Meal 1 (Long Meal with Low Carbohydrate Count) | 76.8 (26.5) | 88.2 (16)
  Meal 2 (Large Meal with Low Carbohydrate Count): number analyzed (Participants) | 14 | 14
  Meal 2 (Large Meal with Low Carbohydrate Count) | 81 (30.8) | 73.7 (33)
  Meal 3 (Small Meal with High Carbohydrate Count): number analyzed (Participants) | 17 | 15
  Meal 3 (Small Meal with High Carbohydrate Count) | 62.7 (20.2) | 59.9 (26.8)
  Meal 4 (Large Drink with No Carbohydrates): number analyzed (Participants) | 16 | 15
  Meal 4 (Large Drink with No Carbohydrates) | 91.9 (14.1) | 84.3 (18.1)
  Meal 5 (Typical Meal Size with Medium Carbohydrate Count): number analyzed (Participants) | 15 | 15
  Meal 5 (Typical Meal Size with Medium Carbohydrate Count) | 91.8 (10.8) | 76.4 (26.9)
  Meal 6 (Long Meal with High Carbohydrates): number analyzed (Participants) | 15 | 15
  Meal 6 (Long Meal with High Carbohydrates) | 74.2 (25.9) | 62.8 (33)
  Meal 7 (Large Drink with High Carbohydrate): number analyzed (Participants) | 15 | 15
  Meal 7 (Large Drink with High Carbohydrate) | 74.8 (16.5) | 67.8 (25.6)
  Meal 8 (Typical Meal Size with Low Carbohydrate Count): number analyzed (Participants) | 15 | 15
  Meal 8 (Typical Meal Size with Low Carbohydrate Count) | 86.4 (15.2) | 90.8 (14.2)

ADVERSE EVENTS:
Time Frame: Overall subject participation lasted approximately 3 weeks to 6 months, which included a run-in period and a study period (5 days at-home and 5 days in-clinic).
Groups:
- Phase 1 (Software Release Tag 1.0): Phase 1 studied the Klue Health app with investigational software release tag 1.0
- Phase 2 (Software Release Tag 2.0): Phase 2 studied the Klue Health app with investigational software release tag 2.0
Arm/Group | Phase 1 (Software Release Tag 1.0) | Phase 2 (Software Release Tag 2.0)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/18
Other Adverse Events (participants affected / at risk) | 1/18 | 1/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (Software Release Tag 1.0) (N=18) | Phase 2 (Software Release Tag 2.0) (N=18)
Severe Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (Software Release Tag 1.0) (N=18) | Phase 2 (Software Release Tag 2.0) (N=18)
Indigestion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/28/NCT04964128/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT04964128/SAP_001.pdf